CLINICAL TRIAL: NCT06542354
Title: Effect of Prehabilitation on Rectal Cancer Surgery Following Neoadjuvant Chemoradiotherapy: A Randomized Prospective Cohort Study
Brief Title: Prehabilitation During Neoadjuvant Chemoradiotherapy for Rectal Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xu jianmin, Professor, Fudan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: preHab-rectal
Record Dates: First submitted 2022-01-17; First posted 2024-08-07 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Rectal Cancer
Keywords: prehabilitation
MeSH Terms: conditions — Rectal Neoplasms | interventions — Exercise

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prehabilitation (Experimental): 6-week trimodel prehabilitation program consists of physical exercises, nutrition supplement and mental support for patients with rectal cancer during neoadjuvant chemotherapy before surgery. All patients will receive ERAS care pattern after surgery.
  Interventions: Behavioral: Physical exercise; Dietary Supplement: Nutrition supplement; Behavioral: Mental support
- Standard care (No Intervention): Patients receive no specific interventions mentioned above during their neoadjuvant chemoradiotherapy. All patients undergoing primary leision resection will receive postoperative ERAS care.

INTERVENTIONS:
Behavioral: Physical exercise — Physical exercises personally scheduled consisting of daily aerobic exercise(30mins) of fast walking(≥5km) and resisitance training.
  Arms: Prehabilitation
Dietary Supplement: Nutrition supplement — Nutritional counselling is given to patients to ensure their daily proteins and energy requirements are met. Oral nutrition supplement (ENSURE) is provided daily seperated in 2 doses
  Arms: Prehabilitation
Behavioral: Mental support — Relaxation exercise and psychological counselling delivered by weekly telephone follow-up
  Arms: Prehabilitation

SUMMARY:
The purpose of this study is determine whether a trimodel prehabilitation program (combined with physical exercise, nutrition supplement and mental support) during neoadjuvant chemoradiotherapy can help patients with rectal cancer to achieve better postoperative outcomes include perioperative complication rate, functional outcomes and quality of life.

DETAILED DESCRIPTION:
This study is a prospective, single-center, randomized control trial. Including criteria were (1) Age between 18 and 80 years; (2) Histologically confirmed rectal adenocarcinoma；(3) Performance status (ECOG) 0-2; (4) Undergoing/scheduled for neoadjuvant chemoradiotherapy lasting at least 4 weeks. (5) Fried frailty score ≥2. Patients operated as emergency, pregnant or with comodities constraining physical exercise or causing disturbance of consciousness are excluded.

All particapants were recruited and randomly assigned to receive trimodel prehabilitation program or standard care. All patients were treated with an ERAS protocol. The primary end-point is postoperative complications within 30 days. Complications were diagnosed and classified according to the Clavien-Dindo classification and comprehensive complication index was calculated. The secondary end-points were functional walking capacity, hospital length of stay, nutrition status, patient-reported health related quality of life and immune function markers. The study was approved by the Ethics Committee of Zhongshan Hospital, Fudan University, Shanghai, China. Written informed consent was obtained for patients to participate the study. This study followed the Consolidated Standards of Reporting Trials (CONSORT) reporting guideline.

ELIGIBILITY:
Inclusion Criteria:

* Patients with rectal cancer undergoing/scheduled for neoadjuvant chemoradiotherapy
* Fried Frailty score≥2 (intermediately frail or frail)
* Written consent informed

Exclusion Criteria:

* Co-morbiditie contraindicating physical exercise or causing disturbances of conciousness (dementia, Parkinson Disease, previous stroke with paresis, taking carbidopa/levodopa, donepezil or antidepressants)
* Emergent surgery
* ASA grade IV-V
* Pregnancy (absence confirmed by serum/urine β-HCG) or breast-feeding
* Known drug abuse/ alcohol abuse

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2021-12-20 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2024-03-20 (Actual)

PRIMARY OUTCOMES:
Functional outcome | at baseline, before surgery, 4 weeks and 8 weeks after surgery
  Walking capacity measured by 6-minute walking distance (6MWD)

SECONDARY OUTCOMES:
perioperative complication | recorded from the day of surgery to 30 days after surgery
  measured by comprehensive complication index (CCI)
Nutrition status | at baseline, before surgery, 4 and 8 weeks after discharge
  measured by BMI and SMI
Patient-reported outcome measures | at baseline, before surgery and 30days after discharge
  using SF-36
immune function markers | at baseline, before surgery, 4 and 8 weeks after discharge
  specific immnue cells like CD4/CD8, cytokines, peripheral blood test.

CONTACTS AND LOCATIONS:
Overall Officials: Xu Jianmin, MD, Study Director — Fudan University
Locations (1):
- Zhongshan Hospital Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No